CLINICAL TRIAL: NCT05131828
Title: CCMR Two: A Phase IIa, Randomised, Double-blind, Placebo-controlled Trial of the Ability of the Combination of Metformin and Clemastine to Promote Remyelination in People With Relapsing-remitting Multiple Sclerosis Already on Disease-modifying Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Nicholas Cunniffe, Academic Clinical Lecturer, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCTU0269
Record Dates: First submitted 2021-11-12; First posted 2021-11-23 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Metformin; Clemastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Research arm: metformin and clemastine (Experimental)
  Interventions: Drug: Metformin and clemastine in combination
- Control arm: placebos for both metformin + clemastine (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin and clemastine in combination — Metformin hydrochloride 500 mg prolonged release (SR) tablet for oral administration.
  Clemastine hydrogen fumarate 1.34 mg tablet for oral administration.
  Arms: Research arm: metformin and clemastine
Drug: Placebo — Placebo tablets to match both metformin and clemastine tablets.
  Arms: Control arm: placebos for both metformin + clemastine

SUMMARY:
The greatest unmet need for people with multiple sclerosis is an effective therapy for the progressive phase. Current treatments suppress the damage caused by the immune system but there is only a limited window in which these can work. Consequently, much of the research community is turning its attention to the process of repair, called remyelination, in which the lining of nerve cells is reformed. This protects nerves from dying and therefore can delay, prevent, or even reverse, disability progression.

It has previously been shown that stem cells are already present in the brain that can carry out this process. Clemastine, an anti-histamine drug, can instruct them to become active and has already shown a beneficial effect in a phase 2 trial. Now, more recent experiments have shown that changes take place within these stem cells as they age, which prevents them responding to drugs like clemastine, but that this can be reversed by treatment with metformin, a commonly used anti-diabetes drug.

Our goal is to establish whether the combination of metformin and clemastine can promote remyelination in people with MS. We will focus on people with relapsing MS as they will have a greater proportion of nerves healthy enough to allow remyelination to take place, which will maximise the chance of detecting an effect with a smaller sample size.

Participants will also continue treatment with a current disease-modifying MS treatment, to reduce the chance of developing new areas of damage, allowing the trial to focus on the repair process. The treatment duration will be 24 weeks, but given the established safety of the proposed medications, we are able to limit the number of visits to the trial centre to ensure participation is not overly burdensome.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give written informed consent for participation in the trial;
* Male or female, aged between 25 and 50 years (inclusive) at time of signing informed consent form (ICF);
* Relapsing-remitting multiple sclerosis as per the McDonald 2017 criteria (Thompson et al., 2018), including an MRI brain satisfying the McDonald 2017 criteria;
* VEP P100 latency in at least one eye of ≥118 ms;
* Kurtzke EDSS 0.0-6.0;
* At the time of screening being treated with a stable dose for at least 6 months of a category 1 multiple sclerosis DMT or for at least 2 years with a category 2 DMT;
* Able (in the Investigator's opinion) and willing to comply with all trial requirements.

Exclusion Criteria:

* Female participants who are pregnant, lactating or planning pregnancy during the course of the trial;
* Female participants of child-bearing potential whom are unwilling or unable to use one highly effective method of contraception during the trial (as outlined in section 11.11). For the purpose of this document, a woman is considered of childbearing potential, i.e. fertile, following menarche and until post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause;
* Male participants who are unwilling or unable to use contraception during and for 3 months after the trial;
* Participants whom have received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 4 weeks before the screening assessment or is currently enrolled in an interventional investigational trial;
* Retinal nerve layer thickness on spectral-domain optical coherence tomography (OCT) <70 μm in the qualifying eye;
* A clinical episode of optic neuritis in the qualifying eye within the 2 years preceding screening;
* Any unlicensed treatment of multiple sclerosis;
* Any concomitant use of oxybutynin, monoamine oxidase inhibitors (MAOIs), hypnotics or high-dose opiates at screening;
* Significant renal impairment (eGFR <60 mL/min/1.73 m2);
* Screening liver function (alanine aminotransferase, ALT) value greater than 3 times the upper limit of normal;
* Known hypersensitivity to metformin or clemastine (or other arylalkylamine antihistamines) or any of the excipients of these products;
* People taking medication for Diabetes Mellitus at screening;
* People with a diagnosis of epilepsy;
* People with rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption;
* Concurrent use of 4-aminopyridine or fampridine;
* Known contraindication(s) to MRI scanning procedures;
* History of prostatic hypertrophy;
* History of major ophthalmologic disease or concomitant ophthalmologic disorders including glaucoma, macular degeneration, and severe myopia (>-7 Diopters);
* History of stenosing peptic ulcer or pyloroduodenal ulceration;
* History of significant cardiac conduction block or decompensated heart failure;
* History of acute porphyria;
* People with a history of alcohol or other recreational drug misuse within the 6 months preceding screening;
* People unable to avoid alcohol drinks for the course of the trial;
* Vitamin B12 deficiency as defined as B12 levels of < 150 pg/ml measured at screening;
* Any other significant disease, disability or investigation result which, in the opinion of the Investigator, may either put the participant at risk, or may influence the result of the trial, or the participant's ability to participate in the trial.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
the change in the P100 latency of the full-field visual evoked potential (VEP) between baseline and week 26 for each affected eye of participants | Baseline to week 26

SECONDARY OUTCOMES:
The change in MF-VEP latency, between baseline and week 26, for those eyes with delayed latency at baseline | Baseline to week 26
The change in lesional MTR, between baseline and week 26, for the lesions stratified by location | Baseline to week 26
The change in lesional MTR between baseline and week 26, for the lesions stratified by tissue-specific cohort baseline lesional MTR values | Baseline to week 26
Adverse events and withdrawals attributable to metformin and/or clemastine | Baseline to week 28

OTHER OUTCOMES:
The change, between baseline and week 26, in the N75 and N145 latencies of the full-field VEP | Baseline to week 26
The change in full field VEP amplitude, between baseline and week 26, for those eyes with delayed latency at baseline | Baseline to week 26
The change in MF-VEP amplitude, between baseline and week 26, for those eyes with delayed latency at baseline | Baseline to week 26
The change in the number of letters read (and the corresponding LogMAR score) on the Sloan 100%, 2.5% and 1.25% acuity charts, between baseline and week 28 | Baseline to week 28
The change in colour vision between baseline and week 28 | Baseline to week 28
The change in visual fields between baseline and week 28 | Baseline to week 28
The change in saccadic latency parameters in the step, antisaccade and Wheeless tasks between screening and week 28 | Screening to week 28
The change in retinal nerve fibre layer thickness between screening and week 28 | Screening to week 28
The change in MTR of lesional subcomponents and lesional voxels, stratified by location, between baseline and week 26 | Baseline to week 26
The change in lesional MTR between baseline and week 26, for different lesion types | Baseline to week 26
The change in MRI T2 lesion load between baseline and week 26 | Baseline to week 26
The change between baseline and week 26 measured by different MRI biomarkers of remyelination | Baseline to week 26
The change in EDSS between screening and week 26 | Screening to week 26

CONTACTS AND LOCATIONS:
Overall Officials: Nick Cunniffe, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust & University of Cambridge
Locations (1):
- Addenbrooke's Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riboni-Verri G, McMurran CE, Mukherjee T, Daruwalla C, Holland J, Gautam R, Chen BS, Cutting E, Qian W, MacManus D, Chard DT, Brown JWL, Coles AJ, Cunniffe NG. The Cambridge Centre for Myelin Repair trial Two (CCMR Two): a trial protocol for a phase 2a, randomised, double-blind, placebo-controlled clinical trial of the ability of the combination of metformin and clemastine to promote remyelination in people with relapsing-remitting multiple sclerosis already on disease-modifying therapy. Trials. 2025 Dec 8;26(1):562. doi: 10.1186/s13063-025-09254-2. PMID 41361285